#### HONG KONG METROPOLITAN UNIVERSITY

## **Information Sheet**

## TITLE OF THE STUDY

Effects of High-Intensity Focused Electromagnetic Therapy with Pelvic Floor Muscle Training on Urine Leakage and Quality of Life in Primipara or Multipara Women with Stress Urinary Incontinence: A Pilot for Randomized Controlled Trial

## INTRODUCTORY SENTENCE

You are invited to participate in a research study conducted by Hong Kong Metropolitan University Physiotherapy Centre.

## **PURPOSE OF THE STUDY**

This study aims to evaluate the impact of High-Intensity Focused Electromagnetic Therapy (HIFEM) combined with Pelvic Floor Muscle Training (PFMT) versus PFMT alone on urine leakage and quality of life in Primipara or Multipara women with stress urinary incontinence.

## **PROCEDURES**

In this study, you will be randomly assigned to either the experimental group or the control group. The experimental group will receive both HIFEM and PFMT, while the control group will receive only PFMT; the treatment will continue for 6 weeks.

You will also undergo several assessments before and after the 6-week intervention. The measurements will include the 1-hour Pad Test, the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF), and sonography to assess bladder neck movement.

All measurements and interventions are non-invasive.

# POTENTIAL RISKS/STRESS/PAIN/DISCOMFORTS/OTHER FACTORS AND THEIR MINIMIZATION

There will be no direct risks, stress, pain, or discomforts associated with participating in this study.

## POTENTIAL BENEFITS

Participants will receive free treatment from participating in this study.

## PARTICIPATION AND WITHDRAWAL

You have the right to withdraw from the study before or during the measurement without any penalty.

## **CONFIDENTIALITY**

Your personal information and data will not be disclosed to anyone outside the research team. Your name or photo will not appear in any published materials.

## **QUESTIONS AND CONCERNS**

If you have any questions or concerns about the research study, please feel free to contact Prof. William Tsang of HKMU at 3970 8703. If you have questions about your rights as a participant in this research study, please contact the Research Ethics Committee of HKMU at 2768 6251.

## **Consent Form**

# Hong Kong Metropolitan University School of Nursing and Health Studies, Department of Physiotherapy

## **Consent form for**

Effects of High-Intensity Focused Electromagnetic Therapy with Pelvic Floor Muscle Training on Urine Leakage and Quality of Life in Primipara or Multipara Women with Stress Urinary Incontinence: A Pilot for Randomized Controlled Trial

| I have read and understand participate in this study. | the information prov | ided about | the above | study. I | agree | to |
|---|---|---|---|---|---|---|
| Name of participant | Signature of participa | nt | Date | | | |
| Nama of investigator | Signatura of investiga | | Doto | | | |
| Name of investigator | Signature of investiga | WI | Date | | | |